CLINICAL TRIAL: NCT07393347
Title: Pain Neuroscience Education for the Management of Chronic Pain in Elite Volleyball Players With Chronic Shoulder Pain: A Randomized Controlled Trial
Brief Title: Pain Neuroscience Education for the Management of Chronic Pain in Elite Volleyball Players With Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Aziz DENGİZ, Assist. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: valleybollPNE
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Sport Injuries; Volleyball Player
Keywords: pain neuroscience education; volleybal player; shoulder pain
MeSH Terms: conditions — Agnosia; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group randomized controlled design. Eligible participants were randomly allocated to either the pain neuroscience education (PNE) group or the control group. Both groups continued their regular sports training programs, while the intervention group additionally received a structured six-week PNE program. Outcome measures were assessed at baseline and after completion of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience group (Experimental): Participants assigned to this arm received pain neuroscience education (PNE) in addition to their regular sports training program. The PNE intervention was delivered over six weeks, with two sessions per week, each lasting approximately 45 minutes, and focused on the neurobiology and neurophysiology of pain, pain mechanisms, and the relationship between pain and tissue damage.
  Interventions: Other: Pain neuroscience education
- Control group (No Intervention): Participants in the control group continued their regular sports training programs throughout the study period and did not receive pain neuroscience education or any additional educational or therapeutic intervention related to pain management.

INTERVENTIONS:
Other: Pain neuroscience education — Pain Neuroscience Education is an educational intervention aimed at improving individuals' understanding of the neurophysiological mechanisms underlying pain. The education focuses on contemporary pain science concepts, including the role of the central nervous system, pain modulation, central sensitization, and the distinction between tissue damage and pain perception.
  The PNE program was delivered through structured sessions using verbal explanations, visual materials, metaphors, and examples relevant to daily life and sports activities. The content emphasized that pain is a protective output of the nervous system rather than a direct indicator of tissue injury, and that psychological, cognitive, and contextual factors can influence pain intensity and persistence.
  Participants were encouraged to reconceptualize pain, reduce maladaptive beliefs and fear related to movement, and develop a more adaptive understanding of their pain experience. The education was tailored to elite volley
  Arms: Pain Neuroscience group

SUMMARY:
This randomized controlled study investigated the effects of pain neuroscience education (PNE) on pain intensity, pain knowledge, and pain catastrophizing in elite volleyball players with chronic shoulder pain. Participants were assigned to either a PNE group or a control group, both continuing regular sports training, while the PNE group additionally received six weeks of structured education sessions.

DETAILED DESCRIPTION:
This study represents a theory-informed intervention examining chronic shoulder pain in elite athletes from a modern pain science perspective. Instead of focusing solely on peripheral tissue pathology, the research is grounded in the biopsychosocial model of pain, emphasizing the role of central pain processing, pain beliefs, and maladaptive cognitive responses such as catastrophizing. In high-level volleyball players, where repetitive overhead loading and performance demands often lead athletes to continue training despite persistent symptoms, pain may become strongly influenced by cognitive and educational factors. Within this context, the study investigates whether modifying the understanding and interpretation of pain through Pain Neuroscience Education (PNE) can influence both the sensory and cognitive dimensions of the pain experience.

Methodologically, the study was designed as a prospective randomized controlled trial. Elite volleyball players with chronic shoulder pain were randomly allocated to either an education-based intervention group or a control group. Both groups maintained their regular sports training routines, ensuring that any observed effects could be attributed to the educational intervention rather than changes in physical load. The intervention consisted of a structured six-week PNE program delivered in repeated sessions, focusing on explaining pain mechanisms, central sensitization, and the non-linear relationship between tissue damage and pain. Outcomes were selected to reflect both physical and cognitive domains of pain: pain intensity, pain-related knowledge, and pain catastrophizing were measured before and after the intervention period to evaluate multidimensional changes associated with the educational approach.

ELIGIBILITY:
Inclusion Criteria:

* Being an elite volleyball player actively competing in a professional club
* Experiencing shoulder and/or arm pain for at least three months
* Providing voluntary informed consent to participate in the study

Exclusion Criteria:

* Participating in volleyball at an amateur level
* Presence of pain in regions other than the shoulder and arm
* History of cancer or pregnancy
* Pain originating from neurological, cardiogenic, or rheumatological conditions
* Failure to complete the pain neuroscience education (PNE) program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | From enrollment to the end of treatment at 6 weeks"
  The Visual Analog Scale is a unidimensional tool used to assess pain intensity. Participants rate their perceived pain by marking a point on a 10-cm (or 100-mm) horizontal line, with higher scores indicating greater pain intensity.
Revised Pain Neurophysiology Questionnaire (R-PNQ) | From enrollment to the end of treatment at 6 weeks
  Revised Pain Neurophysiology Questionnaire (R-PNQ)
  The R-PNQ is a 12-item questionnaire designed to assess individuals' knowledge of the biology and physiology of pain based on contemporary pain science. Each item is answered as true, false, or undecided. Correct responses are scored as one point, yielding a total score ranging from 0 to 12, with higher scores indicating greater pain neurophysiology knowledge. A validated Turkish version of the questionnaire was used.
Pain Catastrophizing Scale (PCS) | From enrollment to the end of treatment at 6 weeks
  The PCS is a 13-item self-report questionnaire used to evaluate maladaptive cognitive and emotional responses to pain. It consists of three subscales: rumination, magnification, and helplessness. Higher scores reflect greater levels of pain catastrophizing

CONTACTS AND LOCATIONS:
Overall Officials: Aziz DENGİZ, Assist. Prof., Principal Investigator — Muş Alparslan University; Harun KOÇ, Assist. Prof., Study Director — Muş Alparslan University
Locations (1):
- Muş Alparslan University, Faculty of Sport Sciences, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sullivan MJ, Bishop SR, Pivik J. Pain catastrophizing scale. Psychol Assess. 1995;7(4):524-532.
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain. Arthritis Care Res. 2011;63(S11):S240-S252.
- [Background] Catley MJ, O'Connell NE, Moseley GL. Neurophysiology of Pain Questionnaire Rasch analysis. J Pain. 2013;14(8):818-827.
- [Background] Sastre-Munar A, Romero-Franco N. Pain education in youth athletes. Healthcare. 2024;12(2):215.
- [Background] Sánchez-Robalino A, Sinchi-Sinchi H, Ramírez A. Effectiveness of pain neuroscience education in physical therapy: a systematic review and meta-analysis. Brain Sci. 2025;15(6):658.
- [Background] Cuenca-Martínez F, Suso-Martí L, Calatayud J, Ferrer-Sargues FJ, Muñoz-Alarcos V, Alba-Quesada P, et al. Pain neuroscience education in patients with chronic musculoskeletal pain: an umbrella review. Front Neurosci. 2023;17:1272068.
- [Background] Gajardo-Burgos R, Valdebenito-Tejos C, Gálvez-García G, Bascour-Sandoval C. Pain and psychological readiness to return to sport in elite volleyball players. Int J Environ Res Public Health. 2023;20(3):2492.
- [Background] 2. Alaiti RK, Reis FJ. Pain in athletes: current knowledge and challenges. Int J Sports Phys Ther. 2022;17(6):981.
- [Background] 1. Malfliet A, Leysen L, Pas R, Kuppens K, Nijs J, Van Wilgen P, et al. Modern pain neuroscience in clinical practice: applied to post-cancer, paediatric and sports-related pain. Braz J Phys Ther. 2017;21(4):225-232.